CLINICAL TRIAL: NCT01010633
Title: Loteprednol Etabonate Versus Vehicle for the Treatment of Inflammation and Pain Following Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 576
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Results first posted 2012-01-09 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2011-12

CONDITIONS: Inflammation; Pain
MeSH Terms: conditions — Inflammation; Pain | interventions — Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loteprednol Etabonate (Experimental): Loteprednol etabonate
  Interventions: Drug: Loteprednol Etabonate
- Vehicle (Placebo Comparator): Vehicle of loteprednol etabonate
  Interventions: Drug: Vehicle of Loteprednol Etabonate

INTERVENTIONS:
Drug: Vehicle of Loteprednol Etabonate — 1 to 2 drops of vehicle administered into the study eye, 4 times a day for approximately 14 days.
  Arms: Vehicle
Drug: Loteprednol Etabonate — 1 to 2 drops of study drug administered into the study eye, 4 times a day for approximately 14 days.
  Arms: Loteprednol Etabonate

SUMMARY:
This study is being conducted to compare the safety and efficacy of loteprednol etabonate compared to vehicle for the treatment of postoperative inflammation and pain following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are at least 18 years of age.
* Subjects who are candidates for routine, uncomplicated cataract surgery.
* Subjects who, in the Investigator's opinion, have potential postoperative pinholed Snellen visual acuity (VA) of at least 20/200 in the study eye.

Exclusion Criteria:

* Subjects who have known hypersensitivity or contraindication to the study drug or components.
* Subjects with a severe/serious ocular condition, or any other unstable medical condition, that in the investigator's opinion may preclude study treatment or follow-up.
* Subjects with elevated intraocular pressure (>/= 21mm Hg), uncontrolled glaucoma, or being treated for glaucoma in the study eye.
* Subjects who are monocular or have pinholed Snellen VA 20/200 or worse in the non-study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Trusso, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Inc., Rochester, New York, United States

REFERENCES:
- [Derived] Rajpal RK, Fong R, Comstock TL. Loteprednol etabonate ophthalmic gel 0.5% following cataract surgery: integrated analysis of two clinical studies. Adv Ther. 2013 Oct;30(10):907-23. doi: 10.1007/s12325-013-0059-7. Epub 2013 Oct 18. PMID 24136301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was initiated at 20 clinics in the United States (US). Three sites did not enroll any participants. The study was conducted at the remaining 17 sites. First participant was enrolled 11/23/2009 and last participant completed 6/25/2010.
Pre-assignment Details: 406 participants eligible for cataract surgery were enrolled in the study (safety population). 397 participants completed the study.
Groups:
- Loteprednol: Loteprednol etabonate 0.5%
Period: Overall Study
Arm/Group | Loteprednol | Vehicle
Started | 203 | 203
Completed | 199 | 198
Not Completed | 4 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Investigator decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loteprednol | Vehicle | Total
Number analyzed (Participants) | 203 | 203 | 406
Age Continuous [Mean (Standard Deviation); unit: years] | 69.3 (8.73) | 69.0 (9.80) | 69.1 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 122 | 231
  Male | 94 | 81 | 175
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 20 | 16 | 36
  White | 176 | 182 | 358
  Other | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Resolution of Anterior Chamber Cells (ACC).
Description: Number of Study eyes with complete resolution(Grade 0) of anterior chamber cells (ACC) for loteprednol and vehicle. Accumulation of white cells in aqueous graded on a scale of 0-4 where grade 0=no cells. Investigators assessed ACC using a slit lamp.
Time Frame: Visit 5 (Postoperative day 8)
Population: Intent to treat (ITT) population
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Loteprednol | Vehicle
Number analyzed (Participants) | 203 | 203
Number analyzed (Eyes) | 203 | 203
Eyes | 62 | 33
Statistical Analysis 1: Comparison: Loteprednol vs Vehicle; Test type: Superiority or Other; p < 0.001, Chi-squared; Mean Difference (Final Values) = 14.3, 95% CI 2-sided [5.7 to 22.9]

2. Secondary Outcome: Resolution of Anterior Chamber Cells.
Description: Study eyes with complete resolution of anterior chamber cells (ACC)
Time Frame: At visits 4-7- postoperative day 3, 8,15 & 18
Measure: Number; unit: Eyes
Arm/Group | Loteprednol | Vehicle
Number analyzed (Participants) | 203 | 203
Eyes
  Visit 4 | 17 | 11
  Visit 5 | 62 | 33
  Visit 6 | 102 | 44
  Visit 7 | 96 | 45

3. Primary Outcome: Grade 0 Pain
Description: Number of eyes with grade 0 ocular pain. Ocular pain, defined as a positive sensation of the eye, based on a 0-5 scale where grade 0 equaled no pain and grade 5 equaled severe pain. Ocular pain graded by participants.
Time Frame: Visit 5 (Postoperative Day 8)
Population: Intent to treat population (ITT)
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Loteprednol | Vehicle
Number analyzed (Participants) | 203 | 203
Number analyzed (Eyes) | 203 | 203
Eyes | 148 | 85
Statistical Analysis 1: Comparison: Loteprednol vs Vehicle; Test type: Superiority or Other; p < 0.001, Chi-squared; Mean Difference (Final Values) = 31.0, 95% CI 2-sided [21.4 to 40.7]

ADVERSE EVENTS:
Time Frame: Visit 3 post-operative day 1 thru visit 7 postoperative day 18
Arm/Group | Loteprednol | Vehicle
Serious Adverse Events (participants affected / at risk) | 1/203 | 2/203
Other Adverse Events (participants affected / at risk) | 0/203 | 0/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loteprednol (N=203) | Vehicle (N=203)
Cystoid Macular Edema (Eye disorders) | 1 (1) | 1 (1) — Unrelated to study drug, but probably related to study procedure
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — The event is serious, unexpected, unrelated to the study drug and the study procedure but rather possibly related to a concomitant illness in a predisposed patient
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1) — SAEs were unrelated to study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data generated as a result of this study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee and the Investigator(s) are completed. The results of the study may be published or presented by the Investigator(s)after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.